CLINICAL TRIAL: NCT01948778
Title: The Effects of a Polyethyleneimine-coated Membrane (oXiris™) for Hemofiltration Versus Polymyxin B- Immobilized Fibre Column (Toraymyxin™) for Hemoperfusion on Endotoxin Activity and Inflammatory Conditions in Septic Shock- A Randomized Controlled Pilot Study
Brief Title: The Effects of a Polyethyleneimine-coated Membrane (oXiris™) for Hemofiltration Versus Polymyxin B- Immobilized Fibre Column (Toraymyxin™) for Hemoperfusion on Endotoxin Activity and Inflammatory Conditions in Septic Shock- A Randomized Controlled Pilot Study (ENDoX-study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDoX_CH012
Record Dates: First submitted 2013-08-30; First posted 2013-09-24 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Patients in Septic Shock

ARMS (3):
- oXiris™ filter (Experimental): oXiris™ filter
  Interventions: Device: oXiris™ filter
- Toraymyxin Filter (Experimental): Toraymyxin Filter
  Interventions: Device: Toraymyxin Filter
- Standard of Care (Other): Standard of Care CRRT if necessary
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: oXiris™ filter
  Arms: oXiris™ filter
Device: Toraymyxin Filter
  Arms: Toraymyxin Filter
Device: Standard of Care
  Arms: Standard of Care

SUMMARY:
Septic shock has a high mortality risk despite the availability of various treatments. Endotoxin, that is present in the cell walls of gram-negative bacteria, is a potent trigger of innate immunity. Endotoxin leads to an activation of a cascade with an overwhelming systemic overflow of pro- and anti- inflammatory mediators at the early phase of sepsis with generalized vascular endothelial damage, tissue injury and multi-organ failure.

Extracorporeal blood purification therapies aim to reduce the circulating level of endotoxin. Different extracorporeal blood purification systems are available. The oXiris™ device comprises a surface treated AN69 membrane capable to adsorb a large spectrum of plasma cytokines, such as IL-6 and HMGB1 protein. The positively charged inner surface of the membrane allows absorbing negatively charged bacterial products such as endotoxin. From an historical perspective, filters containing AN69-based membranes have been the most commonly used products for CRRT in the management of critically ill patients and a substantial volume of published data exist.

Another extracorporeal endotoxin removal therapy is the hemoperfusion with ToraymyxinTM (PMX) filter, which is a cartridge selectively removing blood endotoxin. PMX is composed of polymyxin B covalently bonded to polystyrene-derivative fibres. It is well known that the polarity of the polymyxin B antibiotic binds endotoxin and has bactericidal activity. Therefore, the rationale underlying extracorporeal therapy with PMX is to remove circulating endotoxin by adsorption.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria: • Patients with septic shock, defined as 30ml/kg of i.v. fluid administered within a period of 6 hours after initiation of vasopressor therapy with a vasopressor index =3, and at least one of the following criteria: metabolic acidosis, neurologic dysfunction, renal dysfunction, or acute hepatic dysfunction

* Male and Female patients =18 years
* Endotoxin levels =0.6 IU EAA (measured at ICU admission and repeated 24 hours later in case the initial value is =0.4 and <0.6)

Exclusion criteria: • Endotoxin levels <0.6 IU EAA

* Pregnancy or breast feeding
* Neutropenia (circulating neutrophils <500/µl)
* Pre-existing immune deficiencies or immune-suppressive therapy, especially corticosteroids
* Use of Vasopressin (Pitressin?)
* Organ transplantation within the last 12 months
* Terminally ill patients classified as "do not resuscitate"
* History of sensitivity to polymyxin B or to anticoagulant (heparin) HIT or allergy to heparin
* Need for extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2019-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Measurement of the endotoxin activity 72 hours after treatment initiation | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, Prof MD, Principal Investigator — University Hospital Zurich, University Hospital Zurich, Medical intensive care unit
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Derived] Wendel-Garcia PD, Eberle B, Kleinert EM, Hilty MP, Blumenthal S, Spanaus K, Fodor P, Maggiorini M. Effects of enhanced adsorption haemofiltration versus haemoadsorption in severe, refractory septic shock with high levels of endotoxemia: the ENDoX bicentric, randomized, controlled trial. Ann Intensive Care. 2023 Dec 14;13(1):127. doi: 10.1186/s13613-023-01224-8. PMID 38095800
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356